CLINICAL TRIAL: NCT01177943
Title: LY139603 Bioequivalence Study Comparing Atomoxetine Oral Solution and Capsule Formulation in Healthy Adult Male Japanese Subjects
Brief Title: A Bioequivalence (BE) Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 13554; B4Z-JE-LYEO (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Results first posted 2011-10-27 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine Oral Solution (Experimental)
  Interventions: Drug: Atomoxetine
- Atomoxetine Capsule Formulation (Active Comparator)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Administered orally, once.
  Other Names: LY139603; Strattera

SUMMARY:
To demonstrate the bioequivalence of 12.5 milliliters (mL) of atomoxetine oral solution (4 milligrams per milliliter [mg/mL]) compared with 2 capsules of atomoxetine (25 mg per capsule) in healthy adult male Japanese subjects.

ELIGIBILITY:
Inclusion Criteria

* Are healthy Japanese males, as determined by medical history and physical examination
* Have a body mass index (BMI) of greater than or equal to 17.6 and less than or equal to 26.4 kg/m2 at screening
* Cytochrome P450 2D6 (CYP2D6) genotype is categorized as extensive metabolizers (EM) from the result of screening test. EM includes Intermediate Metabolizer (IM) and Ultrarapid Metabolizer (UM).
* Have clinical laboratory test results within normal reference range for the population and investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board governing the site before any trial activities

Exclusion Criteria

* Are investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted.
* Persons who are employed by the sponsor (that is, employees, temporary contract workers, or designees responsible for conducting the study).
* Are currently enrolled in, or discontinued within the last 4 months from, a clinical trial involving an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to atomoxetine (LY139603) or related compounds.
* Are persons who have ever used atomoxetine, or previously participated in this study or any other study investigating atomoxetine and received the study drug.
* An abnormality in the 12-lead ECG that in the opinion of the investigator increases the risk of participating in the study, such as a corrected QT (QTc) interval >450 milliseconds (msec).
* Subjects with a current or past history of clinically significant elevated blood pressure (Supine systolic blood pressure greater than or equal to 140 millimeters of mercury [mmHg] or Supine diastolic blood pressure greater than or equal to 90 mmHg)
* Have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, or metabolism or elimination of drugs or of constituting a risk when taking the study medication or of interfering with the interpretation of data.
* Regularly use known drugs of abuse, or show positive findings on urinary drug screening.
* Have a positive result for Human Immunodeficiency Virus (HIV) test, or show evidence of possible infection.
* Have a positive result for hepatitis B antigen test, or show evidence of possible infection.
* Have a positive result for hepatitis C antibody test, or show evidence of possible infection.
* Have a positive result for syphilis test, or show evidence of possible infection.
* Use or intend to use over-the-counter or prescription medication 7 and 14 days, respectively prior to dosing.
* Blood donation of more than 200 mL of blood and component blood donation within one month prior to dosing, or those who have donated more than 400 mL of blood within 3 month prior to dosing, or history of blood donation of more than 950 mL within the last 12 months.
* Have an average weekly alcohol intake that exceeds 21 units per week or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 360 mL of beer; 150 mL of wine; 45 mL of distilled spirits).
* Subjects with a history of seizure, excluding febrile convulsion in childhood.
* Exposure to a monoamine oxidase inhibitor (MAOI) drug or herbal preparations with central nervous system effects such as St. John's Wort within the last 2 weeks prior to dosing.
* Subjects who have a history or presence of narrow-angle glaucoma.
* Have a history or presence of significant neuropsychiatric disease (for example, maniac-depressive illness, schizophrenia, or depression).
* Currently smoke in excess of 10 cigarettes per day, or equivalent in tobacco or nicotine substitutes, or are unwilling to stop smoking for the duration specified in the protocol
* Subjects determined by the investigator or the sponsor to be inadequate for inclusion in this study for any other reasons.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Atomoxetine Oral Solution First, Then Capsule Formulation: Participants received 50 milligrams (mg) of atomoxetine orally (po), once (12.5 milliliters [mL] at 4 mg/mL). Participants received 2 capsules of atomoxetine (25 mg/capsule po), once.
- Atomoxetine Capsule Formulation First, Then Oral Solution: Participants received 2 capsules of atomoxetine (25 mg/capsule po), once. Participants received 50 mg of atomoxetine po, once (12.5 mL at 4 mg/mL).
Period: First Intervention
Arm/Group | Atomoxetine Oral Solution First, Then Capsule Formulation | Atomoxetine Capsule Formulation First, Then Oral Solution
Started | 21 | 21
Completed | 19 | 21
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Second Intervention
Arm/Group | Atomoxetine Oral Solution First, Then Capsule Formulation | Atomoxetine Capsule Formulation First, Then Oral Solution
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine Oral Solution First, Then Capsule Formulation: Participants received 50 mg of atomoxetine orally (po), once (12.5 mL at 4 mg/mL). Participants received 2 capsules of atomoxetine (25 mg/capsule po), once.
- Atomoxetine Capsule Followed by Oral Solution: Participants received 2 capsules of atomoxetine (25 mg/capsule po), once. Participants received 50 mg of atomoxetine po, once (12.5 mL at 4 mg/mL).
- Total: Total of all reporting groups
Arm/Group | Atomoxetine Oral Solution First, Then Capsule Formulation | Atomoxetine Capsule Followed by Oral Solution | Total
Number analyzed (Participants) | 21 | 21 | 42
Age Continuous [Mean (Standard Deviation); unit: years] | 23.0 (4.4) | 23.4 (2.9) | 23.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 21 | 21 | 42
Race/Ethnicity, Customized [Number; unit: participants]
  Japanese | 21 | 21 | 42
Region of Enrollment [Number; unit: participants]
  Japan | 21 | 21 | 42
weight (kg) [Mean (Standard Deviation); unit: kilograms (kg)] | 62.29 (7.29) | 61.28 (5.90) | 61.79 (6.57)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: The Cmax values are based on the atomoxetine plasma concentration. The Least Squares (LS) Mean Value was based on treatment, period, group, and subject.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 4, 6, 8, 12, 18, and 24 hours post dose
Population: All participants who had a Cmax value were included in the Cmax analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram per millileter (ng/mL)
Groups:
- Atomoxetine Oral Solution: Participants received 50 mg of atomoxetine orally (po), once (12.5 mL at 4 mg/mL).
- Atomoxetine Capsule Formulation: Participants received 2 capsules of atomoxetine (25 mg/capsule po), once.
Arm/Group | Atomoxetine Oral Solution | Atomoxetine Capsule Formulation
Number analyzed (Participants) | 42 | 40
nanogram per millileter (ng/mL) | 456 [420 to 496] | 483 [443 to 526]
Statistical Analysis 1: Comparison: Atomoxetine Oral Solution vs Atomoxetine Capsule Formulation; Test type: Non-Inferiority or Equivalence — 80-125% was used for bioequivalence (BE) criteria in terms of geometric means; ANOVA; Ratio of Geometric LS Mean values = 0.945, 90% CI 2-sided [0.858 to 1.04]

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-tlast)]
Description: The AUC (0-tlast) is the area under the plasma concentration versus time curve from time zero (predose) to time of last quantifiable concentration (tlast) and is based on the atomoxetine plasma concentration. The Least Squares (LS) Mean Value was based on treatment, period, group, and subject.
Time Frame: Predose, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 4, 6, 8, 12, 18, and 24 hours post dose
Population: All participants who had an AUC value were included in the AUC analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: nanogram hour per milliliter (ng*h/mL)
Arm/Group | Atomoxetine Oral Solution | Atomoxetine Capsule Formulation
Number analyzed (Participants) | 42 | 40
nanogram hour per milliliter (ng*h/mL) | 2220 [1950 to 2540] | 2150 [1880 to 2450]
Statistical Analysis 1: Comparison: Atomoxetine Oral Solution vs Atomoxetine Capsule Formulation; Test type: Non-Inferiority or Equivalence — 80-125% was used for bioequivalence (BE) criteria in terms of the ratio of geometric means; ANOVA; Ratio of AUC(0-tlast) values = 1.03, 90% CI 2-sided [1.00 to 1.07]

ADVERSE EVENTS:
Arm/Group | Atomoxetine Oral Solution | Atomoxetine Capsule Formulation
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 9/42 | 6/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine Oral Solution (N=42) | Atomoxetine Capsule Formulation (N=40)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5)
Blood pressure increased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days